CLINICAL TRIAL: NCT04924465
Title: Evaluation of Interstitial Lung Disease Severity in Patients With Antisynthetase Syndrome According to Specific Antisynthetase Antibodies Types
Brief Title: Evaluation of Interstitial Lung Disease Severity in Patients With Antisynthetase Syndrome According to Specific Autoantibodies Profile
Acronym: TYPASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI036
Record Dates: First submitted 2021-05-08; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Antisynthetase Syndrome
Keywords: Interstitial lung disease
MeSH Terms: conditions — Antisynthetase syndrome; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Anti-Jo1: Patients with anti-Jo1 antibodies
  Interventions: Other: Follow-up
- Anti-PL7: Patients with anti-PL7 antibodies
  Interventions: Other: Follow-up
- Anti-PL12: Patients with anti-PL12 antibodies
  Interventions: Other: Follow-up
- Anti-EJ: Patients with anti-EJ antibodies
  Interventions: Other: Follow-up
- Anti-OJ: Patients with anti-OJ antibodies
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Follow-up of clinical data, laboratory tests, radiological data and pulmonary function tests

SUMMARY:
Antisynthetase syndrome (ASS) is an overlap connective tissue disease characterized by the presence of myositis-specific autoantibodies directed against tRNA-synthetases. Clinical manifestations are myositis, interstitial lung disease (ILD), Raynaud's phenomenon, mechanic's hands and polyarthritis. Clinical presentation varies between ASS patients. ASS is potentially life threatening due to lung involvement, especially in rapidly progressive forms. Anti-histidyl-tRNA synthetase (anti-Jo1) antibodies are the most frequently detected antibodies in ASS (60 % of patients). Anti-threonyl-tRNA synthetase (anti-PL7) and alanyl-tRNA synthetase (anti-PL12) antibodies are each detected in 10 % of patients approximatively. Anti-tRNA-synthetases antibodies are mutually exclusive.

Clinical heterogeneity of ASS patients appears to be associated with specific autoantibodies profile. Patients with anti-Jo1 antibodies have a more systemic presentation (especially with muscle involvement), whereas patients with anti-PL7 or anti-PL12 antibodies have more frequent and isolated ILD. If anti-PL7 and anti-PL12 antibodies are associated with more severe ILD and poorer survival is still matter of debate.

Aims of this study were to compare ILD severity at diagnosis and clinical course in patients with ASS according to antisynthetase autoantibodies types.

ELIGIBILITY:
Inclusion Criteria:

* Patients with antisynthetase syndrome according to Connors criteria

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with antisynthetase syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients of rapidly progressive (RP)- ILD | 3 months
  Decrease of at least 10 percent of Forced Vital Capacity (FVC) OR Decrease of at least 5 % of FVC WITH Clinical worsening and/or ILD extension on CT-scan OR Decrease of at least 15 % of Diffusing Capacity of lung for Carbon Monoxide (DLCO) at 3 months of follow-up
Number of patients with severe ILD | Baseline
  Hypoxemia (PaO2 < 60 mmHg) AND/OR Oxygen delivery at time of diagnosis

SECONDARY OUTCOMES:
Number of patients with ILD relapse | 3 years and 5 years
  Clinical worsening AND/OR ILD extension on CT-scan AND/OR Progressive ILD on pulmonary function tests WITH modification of corticosteroids dosage or immunosuppressive drugs during follow-up
Number of patients with chronic respiratory failure | 3 years and 5 years
  Hypoxemia (PaO2 < 70 mmHg) in a stable state during follow-up
Rate of patients without death or lung transplant | 3 years and 5 years